CLINICAL TRIAL: NCT05972707
Title: Magnitude, Types, and Associated Factors of External Abdominal Hernias Among Adult Patients Visiting the Surgical Outpatient Department at Hiwotfana Comprehensive Specialized Hospital and Jugol Regional Hospital, Eastern Ethiopia: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Fufa Miresa, Principal Investigator, Haramaya Unversity
Other Study IDs: Haramaya university
Record Dates: First submitted 2023-07-22; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Abdominal Wall Hernia
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The study was aimed at determining the magnitude, types, and associated factors of external abdominal hernia among adult patients visiting the outpatient department at the Hiwot Fana Comprehensive Specialized Hospital (HFCSH) and Jugol regional hospital in eastern Ethiopia.

DETAILED DESCRIPTION:
A cross-sectional study was carried out from September 20 to December 5, 2022, on adult patients who visited the surgical outpatient department at the Hiwotfana Comprehensive Specialized Hospital and Jugol Regional Hospital in Eastern Ethiopia. All adult patients who visited the surgical outpatient department of each hospital were enrolled in the study using a systematic random sampling technique with skipping intervals of two until the calculated sample size was obtained, which is 403. Data collection was accomplished through medical record reviews of patients and face-to-face interviews. The data were analyzed by the Statistical Package for Social Science version 26 software. Both descriptive and inferential statistics were conducted, and the results were presented in text, graphs, and tables. A Chi-square test was calculated, and an Odds ratio for the strength and directions of association was used with a 95% confidence interval and a P-value of <0.05 to be considered statistical. This investigation determined the overall magnitude of external abdominal wall hernias in the study area as well as the types of external abdominal hernias. At the conclusion of the investigation, each significant associated factor for an external abdominal hernia was identified.

ELIGIBILITY:
Inclusion Criteria:

* All adult individuals who visited the surgical outpatient department during the period of study

Exclusion Criteria:

* Patients who were unable to respond due to severe illness or mental health problems

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult surgical outpatient department patients
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with external abdominal hernia | From September 20, 2022, to December 5, 2022
  Hospital-based magnitudes of external abdominal hernias were studied depending on the identified number of patients with external abdominal hernias.
Types of external abdominal hernias | From September 20, 2022, to December 5, 2022
Associated factors of external abdominal hernias | From September 20, 2022, to December 5, 2022
  The number of participants with external abdominal hernia who have any associated factor for hernia was identified, and the strength of association for each associated factor was determined by using bivariate and multivariate logistic regression studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Haramaya University, Harar, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data sets are to be shared as required to underlie results in a publication.

REFERENCES:
- [Background] CHEUNG LY. Principles of Surgery. Vol. 56, Plastic and Reconstructive Surgery. 1975. 206-207 p.
- [Background] Lassandro F, Iasiello F, Pizza NL, Valente T, Stefano ML, Grassi R, Muto R. Abdominal hernias: Radiological features. World J Gastrointest Endosc. 2011 Jun 16;3(6):110-7. doi: 10.4253/wjge.v3.i6.110. PMID 21860678
- [Background] Qalehsari MQ, Khaghanizadeh M, Ebadi A. Lifelong learning strategies in nursing: A systematic review. Electron Physician. 2017 Oct 25;9(10):5541-5550. doi: 10.19082/5541. eCollection 2017 Oct. PMID 29238496
- [Background] Dabbas N, Adams K, Pearson K, Royle G. Frequency of abdominal wall hernias: is classical teaching out of date? JRSM Short Rep. 2011 Jan 19;2(1):5. doi: 10.1258/shorts.2010.010071. PMID 21286228
- [Background] Muysoms FE, Miserez M, Berrevoet F, Campanelli G, Champault GG, Chelala E, Dietz UA, Eker HH, El Nakadi I, Hauters P, Hidalgo Pascual M, Hoeferlin A, Klinge U, Montgomery A, Simmermacher RK, Simons MP, Smietanski M, Sommeling C, Tollens T, Vierendeels T, Kingsnorth A. Classification of primary and incisional abdominal wall hernias. Hernia. 2009 Aug;13(4):407-14. doi: 10.1007/s10029-009-0518-x. Epub 2009 Jun 3. PMID 19495920
- [Background] Sazhin A, Zolotukhin I, Seliverstov E, Nikishkov A, Shevtsov Y, Andriyashkin A, Tatarintsev A, Kirienko A. Prevalence and risk factors for abdominal wall hernia in the general Russian population. Hernia. 2019 Dec;23(6):1237-1242. doi: 10.1007/s10029-019-01971-3. Epub 2019 May 14. PMID 31089836
- [Background] Rutkow IM. Demographic and socioeconomic aspects of hernia repair in the United States in 2003. Surg Clin North Am. 2003 Oct;83(5):1045-51, v-vi. doi: 10.1016/S0039-6109(03)00132-4. PMID 14533902
- [Background] Groen R, Sesay S, Kushner A, Dumbuya S. Three-stage repair of a giant inguinal hernia in Sierra Leone: A management technique for low-resource settings. J Surg Case Rep. 2011 Dec 1;2011(12):8. doi: 10.1093/jscr/2011.12.8. PMID 24971839
- [Background] Arifin WN. Introduction to sample size calculation. Educ Med J. 2013;5(2):89-96.
- [Background] Kibret AA, Tekle SY, H/Mariam MM, Worede AG, Dessie MA. Prevalence and associated factors of external hernia among adult patients visiting the surgical outpatient department at the University of Gondar Comprehensive Specialised Hospital, Northwest Ethiopia: a cross-sectional study. BMJ Open. 2022 Apr 15;12(4):e056488. doi: 10.1136/bmjopen-2021-056488. PMID 35428635
- [Background] Mahfouz MEM, Al-Juaid RS. Prevalence and risk factors of abdominal hernia among Saudi population. J Family Med Prim Care. 2021 Aug;10(8):3130-3136. doi: 10.4103/jfmpc.jfmpc_622_21. Epub 2021 Aug 27. PMID 34660458
- [Background] Iqbal MN, Akhter S, Irfan M. Prevalence of hernia in relation to various risk factors in Narowal , Pakistan. 2015;3(1):29-32.
- [Background] Rao G, Rao A, Pujara N, Pujara P, Patel S. Prevalence Of Hernia Among Fishermen Population In Kutch District, India -. Natl J Integr Res Med. 2015;6(4):44-51.